CLINICAL TRIAL: NCT07216417
Title: TeleYoga for Chronic Low Back Pain: A Quantitative and Qualitative Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taylor Rees (Other)
Responsible Party: Sponsor-Investigator, Taylor Rees, Sponsor-Investigator, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00161902
Record Dates: First submitted 2025-10-07; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Low Back Pain
Keywords: yoga; mindfulness
MeSH Terms: conditions — Low Back Pain | interventions — Yoga; Mindfulness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga + Mindfulness (Experimental): These participants will synchronously on zoom watch 2 recorded classes with a coach to guide them. Classes are 2x a week for 4 weeks. Their classes will be a mix of physical yoga postures and mindfulness ie meditation and breathing exercises.
  Interventions: Behavioral: Yoga; Behavioral: Mindfulness
- Yoga - Mindfulness (Active Comparator): These participants will synchronously on zoom watch 2 recorded classes with a coach to guide them. Classes are 2x a week for 4 weeks. Their classes will only be physical yoga postures
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — Physical Yoga postures
Behavioral: Mindfulness — breathing cues or meditation practice
  Arms: Yoga + Mindfulness

SUMMARY:
Chronic low back pain (CLBP) is a highly prevalent and debilitating condition, affecting 84% of the population over a lifetime1. CLBP is the leading cause of disability worldwide 2 and is a top condition for health care expenditure in the US3. Emerging evidence indicates that individuals with low back pain have altered neurophysiological processes within the central nervous system leading to high prevalence of anxiety and depression, and poor sleep quality4-7. Standard treatments often focus on the local source of pain; however, for many patients the persistence and severity of pain cannot be explained by peripheral pathology alone. Yoga is a promising mind-body integrative intervention, as it targets the psychological and neurophysiological aspects of pain. The efficacy of yoga practice for reducing pain8,9 and psychological distress10,11 has been shown by many systematic reviews and randomized control trials (RCTs)12-16. Additionally, mindfulness, meditation, and breathwork interventions produce meaningful improvements in pain17,18, anxiety19,20, depression21, and sleep quality22,23.

Evidence clearly indicates yoga is an effective intervention for management of chronic LBP9. However, the majority of prior RCTs have included in-person yoga sessions 24-26, which may be a barrier to many people. Recently, virtual delivery of interventions is gaining popularity. A few recent studies reported promising feasibility of tele-yoga in people with various chronic pain conditions e.g. Alzheimer's 27, dementia 28, and knee osteoarthritis 29. Only one recent RCT conducted tele-yoga intervention for people with CLBP and resulted in decreased pain 14, but is limited to quantitative measures only and did not compare yoga against active therapy. No study has assessed participants' perspective of virtual yoga intervention for chronic low back pain, which is important to determine feasibility of tele-yoga for CLBP management. The objectives of this study are two fold: 1) to investigate the acceptability of yoga intervention using a tele-yoga approach and 2) to compare the effectiveness of a tele-yoga intervention with a mindfulness focus (Y+M) to a tele-yoga intervention without a mindfulness focus (Y-M) in adults with CLBP.

Thirty participants27,30 with CLBP aged 30-8014 will be recruited and randomly assigned to Y+M or time-matched Y-M (physical movement without breathing and meditation) group. Each group will participate in video-guided live group sessions 2x a week for 4 weeks28,30.

Aim 1: To evaluate acceptability of tele-yoga intervention for CLBP. The investigators will assess acceptability via participants' overall satisfaction using 1) self-reported satisfaction ratings, the Acceptability of Intervention Measure (AIM)31 and 2) semi-structured qualitative interviews to capture participant feedback about their experience (e.g. barriers, facilitators, motivators, perceived effectiveness, self-efficacy). Hypothesis 1: Participants will have good acceptability to tele-yoga intervention.

Aim 2: To compare between-group changes in pain and function between tele-yoga with breath regulation, focused attention/meditation and tele-yoga without breath regulation, focused attention/meditation. Efficacy of tele-yoga on pain and function between groups will be assessed at baseline, midpoint, and post-intervention. Pain (VAS) and function (ODI) will serve as primary outcomes. Clinically significant improvement is defined as ODI scores ≥15% and reductions in VAS pain scores ≥2 points as compared to the sham yoga group. Secondary outcomes will include PROMIS Pain Interference Short Form. Hypothesis 2: The Y+M will have greater improvements than the YG.

Aim 3: To compare between-group changes in psychological health between tele-yoga with breath regulation, focused attention/meditation and tele-yoga without breath regulation, focused attention/meditation. Psychological measures include Beck Anxiety Inventory, Beck Depression Inventory, Pittsburg Sleep Quality Index and compared between both groups. Secondary measures include symptoms of CS with standard measures of Fibromyalgia 2016 (FM) survey32. Hypothesis 3: The Y+M will have greater improvements than the Y-M.

This project is highly innovative in its focus on 1) gaining participants' perspective with tele-yoga delivery and 2) telehealth-delivered, mind-body intervention specifically targeting central pain sensitization in CLBP with potential exploration of underlying mechanisms of yoga. The project is significant with potentially improving access to virtual treatment options that may potentially lead to self-management of CLBP. Expected outcomes of this research include evidence to support tele-yoga as an effective, accessible integrative therapy for reducing centrally mediated pain symptoms.

DETAILED DESCRIPTION:
Background and Significance

CLPB is a highly prevalent condition worldwide, affecting approximately 619 million people in 2020 with an estimated projection of impacting 843 million by 20502. In the United States, it is a leading cause of disability and work limitation33 and imposes enormous socioeconomic costs, with U.S. healthcare expenditures for CLBP estimated in the tens of billions of dollars annually (around $40 billion in direct costs)34 and total costs exceeding $100 billion per year35. Beyond its economic burden, CLBP significantly can impair physical function and psychological well-being. CLBP is accompanied with substantial psychological distress, with notably elevated rates of both anxiety and depression36. Individuals with CLBP had almost 5x the prevalence of anxiety or depression as compared to those without pain36. In addition to higher anxiety and depressive scores, CLBP has been associated with poorer physical function, greater limitations in daily activities and lower quality of life, even after adjusting for demographics and comorbidities37.

A subpopulation of CLBP patients exhibits evidence of nervous system hyperactivity characterized by widespread hyperalgesia, amplified pain signaling, and impaired pain modulation38. Studies indicate that this subgroup may comprise a substantial fraction of CLBP cases (with prevalence estimates ranging broadly and averaging around 40-50%)33,39. Clinically, these patients tend to have more severe pain manifestations and are less likely to respond to standard treatments40, highlighting the need for tailored therapeutic approaches. One promising non-pharmacological treatment for CLBP is yoga, a mind-body therapy. Systematic reviews and meta-analyses have found that yoga practice leads to significant improvements in pain intensity and functional disability in CLBP patients41. Yoga has been generally well-tolerated with no serious adverse effects, making it a valuable conservative adjunct in the management of CLBP41.

The delivery of yoga interventions via telehealth ("tele-yoga") has rapidly expanded in recent years, especially during the COVID-19 pandemic, to improve access for individuals with chronic health conditions who may have difficulty attending in-person classes 42. Chronic conditions such as persistent pain, cancer, and neurocognitive disorders can limit mobility and increase barriers to participating in on-site exercise programs. Tele-yoga, defined as live-streamed, interactive yoga instruction via videoconferencing, offers a potential solution by allowing patients to engage in supervised mind-body exercise from home 42,43. Early studies have suggested that remotely delivered yoga is feasible across a range of chronic illnesses 43,44. However, the evidence remains limited, with most studies to date being small pilot trials or program evaluations focused on feasibility and acceptability rather than large efficacy trials 44,45. In addition, many prior remote yoga interventions have used asynchronous (pre-recorded) content, whereas fewer have examined synchronous (real-time) group yoga, which may better replicate the social and therapeutic aspects of in-person classes 44,46.

Mindfulness, meditation, and breathwork interventions produce meaningful improvements in pain17,18, anxiety19,20, depression21, and sleep quality22,23. Mindfulness-based interventions such as Mindfulness-Based Stress Reduction (MBSR) and Mindfulness-Based Cognitive Therapy (MBCT) have been shown to reduce low back pain-related disability and psychological distress, with effects comparable to pharmacologic and cognitive-behavioral therapies47,48 Breathing practices, including slow and structured techniques, similarly improve autonomic regulation and mood18, and meditation-based programs consistently demonstrate moderate improvements in anxiety, depression, and sleep quality. Collectively, these findings highlight the potential of mind-body practices as safe, accessible, and evidence-based approaches to enhance both physical and psychological outcomes.

Patients with chronic conditions and their caregivers have expressed both enthusiasm and concerns regarding online interventions. Convenience, home comfort, and improved access are frequently cited advantages of tele-yoga, while drawbacks include technology challenges, distractions at home, and the absence of hands-on guidance or in-person community support 43. Understanding user perspectives and the outcomes of tele-yoga interventions is essential for determining the role of tele-yoga in chronic disease management. Accordingly, we conducted a systematic review of "TeleYoga for Chronic Conditions" to synthesize the emerging evidence on synchronous tele-yoga interventions for individuals with chronic health conditions. There were only 9 studies that tested tele-yoga to date (manuscript in preparation) that are presented in Table 1 and 2. These studies represent a cross-section of tele-yoga research in chronic pain, cancer survivorship, dementia, and integrated care settings, suggesting current gap related to tele-yoga intervention in CLBP. The investigators additionally draw on related literature for context and discussion, while not duplicating the detailed analysis of any study beyond our scope. Importantly, of the 9 studies, only one study conducted qualitative work. It is important to examine the feasibility of tele-yoga for CLBP management that may potentially facilitate self-management strategies in individuals.

Reviews of literature identify the lack of studies utilizing tele-yoga for CLBP management even though CLBP continues to be reported as the leading cause of disability.

Overall gaps in knowledge:

* There are no studies evaluating qualitative feedback from participants with chronic low back pain being treated with tele-yoga.
* A Recent study14 has looked at utilizing tele yoga to treat CLBP. However, this study only recruited from a single employer health-based health plan and utilized a wait list control instead of an active control.
* Most studies only utilize self-report measures (pain, disability, etc.). One study53 examined central sensitization (CS) subjective information, however did not take all objective measures that are typically associated with central sensitization or pain battery (Quantitative Sensory Testing).

As tele-yoga practice gains traction, it is important to understand participants' perspective of their experiences, barriers, and facilitators to improve implementation of tele-yoga practices.

B. Rationale Our goal is to not only determine the feasibility of tele yoga, but to explore participant feedback that can help further identify barriers to interventions in tele-yoga group session format. By utilizing the stretching intervention as active control group, The investigators will be able to determine the benefit of tele yoga as compared to stretching telehealth intervention. Finally, the investigators plan to give local participants the opportunity to come to KUMC so that the investigators can gather objective data of CS rather than relying solely on self-report data as many other yoga studies have done in previously published literature.

II. Research Plan and Design

A. Study Objectives:

Aim 1: To evaluate acceptability of tele-yoga intervention for CLBP. The investigators will assess acceptability via participants' overall satisfaction using 1) self-reported satisfaction ratings, the Acceptability of Intervention Measure (AIM)31 and 2) semi-structured qualitative interviews to capture participant feedback about their experience (e.g. barriers, facilitators, motivators, perceived effectiveness, self-efficacy). Hypothesis 1: Participants will have good acceptability to tele-yoga intervention.

Aim 2: To compare between-group changes in pain and function between tele-yoga with breath regulation, focused attention/meditation and tele-yoga without breath regulation, focused attention/meditation. Efficacy of tele-yoga on pain and function between groups will be assessed at baseline, midpoint, and post-intervention. Pain with Visual scale analog (VAS) and function with Oswestry Disability Index (ODI) will serve as primary outcomes. Clinically significant improvement is defined as ODI scores ≥15% and reductions in VAS pain scores ≥2 points as compared to the sham yoga group. Secondary outcomes will include PROMIS Pain Interference Short Form. Hypothesis 2: The Y+M will have greater improvements than the YG.

Aim 3: To compare between-group changes in psychological health between tele-yoga with breath regulation, focused attention/meditation and tele-yoga without breath regulation, focused attention/meditation. Psychological measures include Beck Anxiety Inventory, Beck Depression Inventory, Pittsburg Sleep Quality Index and compared between both groups. Secondary measures include symptoms of CS with standard measures of Fibromyalgia 2016 (FM) survey32. Hypothesis 3: The Y+M will have greater improvements than the Y-M.

Primary outcomes:

Acceptability outcomes (Aims 1)

1. Acceptability of Intervention Measure (AIM)31 and semi-structured qualitative interview.
2. Feedback will be obtained via both quantitative and qualitative measures. Quantitatively, participant will be asked to rate how acceptable the intervention yoga for LBP was on a scale from 0 ("Not helpful at all") to 10 ("Extremely helpful"). Qualitative: Semi-structured interviews of the tele-yoga group will be conducted at the completion of the study to capture their feedback about their experience of synchronous tele-yoga group sessions and video-recorded self-practice. Interview will include open-ended questions e.g. what they liked about the intervention, what parts of the intervention where the most/least helpful in addressing their symptoms, how they would change the intervention, whether they had any challenges completing the intervention, and whether they had anything else to share about their time in the study. A current draft of the semi-structured interview guide is provided (Appendix1)

Pain and function outcomes (Aim 2) Oswestry Disability Index54: This is used to gauge function of those with spinal disorders

VAS: Visual analog scale: This is used to measure pain on a 10 point scale PROMIS Pain Interference Short Form55: This is used to assess the extent to which pain interferes with social, cognitive, emotional, and physical activities

Psychological outcomes (Aim 3) Beck Anxiety Index (BAI)56: The BAI is a self-report questionnaire that measures the severity of anxiety. It contains 21 multiple-choice questions; each answer is scored on 0 (not at all) to 3 (severely) scale. Higher scores indicate more severe anxiety symptoms.

Beck Depression Inventory (BDI-I)57. The BDI contains 21-questions with each answer being scored on a scale value of 0 to 3 and higher scores indicating more severe depression symptoms. Scores range from minimal depression (0-13), mild depression (14-19) moderate depression (20-28) and severe depression (<29). A score of ≥ 20 indicates moderate to severe depression and the person would be excluded from participating upon completion of the baseline questionnaire.

Pittsburg Sleep Quality Index (PSQI) 58: This is used to assess sleep quality and disturbances over a one month period. A total PSQI score of >5 indicates poor sleep quality.

2016 FM survey32: This is used to measure widespread pain and co-morbid symptoms. 2011 FM survey will be completed at pre and post sleep-restriction and post recovery period.

B. Study Type and Design: This is a feasibility RCT where participants will be randomized into to Y+M (n=20) versus Y-M (n=20) group. After receiving IRB approval, participants will be recruited from word of mouth, community and social media methods (e.g. broadcast email, the PI's lab page, Facebook, Instagram, etc). Participants will be screened via phone call, RedCap survey or email correspondence.

30 individuals with chronic low back pain (CLBP) will be enrolled in our study. Participants will be asked to fill out general health history, FM 2016, ODI VAS, PROMIS, BAI, BDI, and PSQI questionnaires prior to beginning . Participants will be randomized into either the yoga group or the sham yoga (mobility) group. Yoga intervention and sham yoga intervention will be taught by the same physical therapist who is also a certified yoga instructor. Classes will be recorded and then played during participants live synchronous time. Both groups will complete a 4 week intervention. During the study period they will participate in their intervention for 2x a week for 4 weeks.

Tele-Yoga + M intervention:

Each week the yoga group will follow the same class structure (Check in with participants, Yoga philosophy, Postures and breathing practice, Relaxation, Closing)14. The course will have a different theme each week and progress the physical postures as the participants are able. The physical postures will include poses sitting in a chair (examples: shoulder circles, seated neck stretches, seated pelvic tilts, cat/cow, chair twist, etc), standing behind a chair (example: mountain pose, chair/modified chair pose, modified down dog pose/down dog pose, etc) and laying on the floor (example: bridge/supported bridge pose, knees to chest, open books, cobra, table pose, spinal extension pose, etc). All these poses and activities have been shown to be feasible and effective in management of CLBP. Breathing practices will be incorporated into physical posture for mind-body integration.

Tele-Yoga -M Intervention:

Mobility and Flexibility exercises that are similar to the physical aspects of yoga will be provided to this group. The exercises will include exercises that are very similar/the same as the yoga group: The physical postures will include poses sitting in a chair (examples: shoulder circles, seated neck stretches, seated pelvic tilts, cat/cow, chair twist, etc), standing behind a chair (example: mountain pose, chair/modified chair pose, modified down dog pose/down dog pose, etc) and laying on the floor (example: bridge/supported bridge pose, knees to chest, open books, cobra, table pose, spinal extension pose, etc).

This class will not have any emphasis on breathing, relaxation or yoga philosophy. The entire time will be spent performing total body general mobility and stretching exercises.

Participants in both groups will be asked to report any questions, concerns or increase in pain experience to their instructor as soon as they are able.

The class will be performed on Zoom to ensure KUMC HIPAA compliance.

Study Procedures: The investigators will enroll individuals aged 30-80 years old with CLBP. All participants meeting the inclusion/exclusion criteria will complete a baseline assessment. Once participants have completed redcap baseline assessment material, they can be enrolled. Once enrolled, participants will fill out additional questionnaires. Participants who live a reasonable driving distance to KU, will have the option of coming to campus for objective measure testing. Then, participants will be randomized by the yoga instructor (to blind the rest of the research team) into the yoga group or the time matched stretching group. Both groups will perform live weekly classes and be encouraged to perform the recordings of the live class a minimum of two times per week.

All the methods used in this study are for the purpose of research.

Study design and timeline:

Initial screening and consenting: In this part, the investigators will identify subjects according to the inclusion and exclusion criteria.

Baseline assessment: can occur during consenting or separately as participants desire Mid-term assessment of questionnaires (2 weeks into the study) Final assessment at the completion of the study (4 weeks)

Subject Participation

A. Recruitment:

The investigators will primarily recruit patients via word of mouth, by placing study flyers throughout KU hospital and KUMC and social media e.g. broadcast, facebook, etc. Attach is a copy of study flyer

B. Screening Interview/questionnaire: Screening will be conducted electronically via redcap survey or email or by phone interview, whichever method is preferred by the potential participant. A copy of the screening form is attached.

C. Informed consent process and timing of obtaining of consent

1. Taylor Rees, PT, DPT; Neena Sharma, PT, PhD
2. Initial written consent will be obtained prior to the initial assessment. Informed consent will be done following a detailed review of the screening form by one of the indicated research personnel. Participants will be encouraged to ask questions and research personnel will ask if participants have further questions after answering any questions. The consent interview and assessments will be conducted in a private area in the clinic or in via video call on HIPAA compliant Zoom. If a potential participant declines, they will be thanked for their time. Part of the screening detects which subjects may not be able to provide consent due to potential cognitive impairment or psychological issues, and they will be excluded from the study.
3. Potential participants interested in participating in the study will give their consent. Only adults and English-speaking individuals will be recruited. Based on the screening form, the study team will determine participants' eligibility.

D. Alternatives to Participation: The alternative to participation is to not participate E. Costs to Subjects: There is no financial burden for participants. Questionnaires would be completed in-person or online and provided by the study personnel without any charge.

F. How new information will be conveyed to the study subject and how it will be documented: New information will be conveyed to participants in person or via HIPAA compliant Zoom.

G. Payment, including a prorated plan for payment: Participants will not receive payment.

H. Payment for a research-related injury: There is no payment for research related injury as expressed in informed consent form. This is a minimal risk associated with this study.

IV. Data Collection and Protection

A. Data Management and Security:

Each participant will be assigned a unique de-identified subject code. This number will be placed on the consent form and will correspond with the subject's data sheets and session notes so that only the consent form will contain both the participant's name and code. The consent forms will be kept in a locked filing cabinet in the office of the principal investigator. Data from testing will be stored on a spreadsheet using the unique subject code and stored on a secure network drive (S drive or G drive) with access only provided to the investigator and research assistants. No data forms will contain any specific participant identifiers. All data collected will be evaluated and analyzed only as group data and no specific participants will be identified in presentation or publication of study results.

The consent interview and all assessments will be conducted in a private area in CORR lab or via HIPAA compliant Zoom. Only participants will use the laboratory space assessments. Findings will be available to those participants who express interest at any time upon completion of the study. All research study personnel will complete Human Subjects training, HIPAA Research Training and file a Conflict of Interest Disclosure.

The code will be stored in secure network drive (P drive) with access only provided to the primary investigator and research assistants.

Each participant will be assigned a unique de-identified subject code. This number will be indicated on the consent form and will correspond with the subject's data sheets and session notes so that only the consent form will contain both the participant's name and code.

Mobile devices used for survey outcomes will be linked via a special code to a REDCap survey which will be completed in a de-identified coded manner.

ELIGIBILITY:
Inclusion Criteria:

* 30-80 year old individuals
* Ability to speak, read and write English as needed for study LBP for 3 months with frequency of 2 or more days/week or daily low back pain for the most recent three months
* Pain intensity minimum 3 on 0-10 pain scale where 0=no pain and 10=maximum pain imagined
* Have internet access and device available for logging into virtual yoga classes
* Be able to get on and off the floor

Exclusion Criteria:

* spine compression, tumor, infection, spine surgery within the last 12 months
* neurological conditions such as stroke, Parkinson's disease, Alzheimer's disease or other cognitive impairments.
* pregnancy
* currently performing yoga or has performed yoga on a regular basis within the last 6 months

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Semi Structured Interview | Week 4
  This interview will take about 30-60 minutes, but we can take a break anytime you need to. If you need to end the interview at any time, please let me know and we will stop.
  Do you have any other questions before we start? Are you still willing to continue with this interview? Do you mind if we start the audio-recorder?
  1. I would like to begin this interview by asking you, before you started this project what your experience with yoga was.
     1. [Clarifying probe]: Had you ever practiced yoga before?
     2. [If have practiced before]: Prior to this project what were your main goals for doing yoga? How many times a week were you doing yoga?
     3. [If have not practiced before] What led you to want to take part in this yoga program?
  2. Why did you join a yoga study?:
     1. [Clarifying probe]: Before you started this program, what were you hoping to get out of doing yoga?
     2. [Clarifying probe]: What did you hope doing this yoga program would do for you?
  3. What was your overall experienc
Acceptability of Intervention Measure (AIM) | Week 0, Week 2, Week 4
  Acceptability of Intervention Measure (AIM)
  1. [Triple P/Implementation Strategy] meets my approval.
  2. [Triple P/Implementation Strategy] is appealing to me.
  3. I like [Triple P/Implementation Strategy].
  4. I welcome [Triple P/Implementation Strategy]. Intervention Appropriateness Measure (IAM)
  1) [Triple P/Implementation Strategy] seems fitting. 2) [Triple P/Implementation Strategy] seems suitable. 3) [Triple P/Implementation Strategy] seems applicable. 4) [Triple P/Implementation Strategy] seems like a good match. Feasibility of Intervention Measure (FIM)
  1. [Triple P/Implementation Strategy] seems implementable.
  2. [Triple P/Implementation Strategy] seems possible.
  3. [Triple P/Implementation Strategy] seems doable.
  4. [Triple P/Implementation Strategy] seems easy to use.

SECONDARY OUTCOMES:
Oswestry Disability Index | Week 0, Week 2, Week 4
  Section 1 - Pain intensity I have no pain at the moment The pain is very mild at the moment The pain is moderate at the moment The pain is fairly severe at the moment The pain is very severe at the moment The pain is the worst imaginable at the moment
  Section 2 - Personal care (washing, dressing etc) I can look after myself normally without causing extra pain I can look after myself normally but it causes extra pain It is painful to look after myself and I am slow and careful I need some help but manage most of my personal care I need help every day in most aspects of self-care I do not get dressed, I wash with difficulty and stay in bed
  Section 3 - Lifting I can lift heavy weights without extra pain I can lift heavy weights but it gives extra pain Pain prevents me from lifting heavy weights off the floor, but I can manage if they are conveniently placed eg. on a table Pain prevents me from lifting heavy weights
Promis Short Form | Week 0, Week 2, Week 4
  The PROMIS Pain Short Form are short, reliable surveys that measure how much pain someone has (intensity), how much it gets in the way of life (interference), and sometimes how much it shows on the outside (behavior). They are quick to administer, produce standardized T-scores, and are widely used in clinical trials and practice to monitor pain outcomes.
Visual Analog Scale | Weekly
  Pain rating 0-10 at current, best, worst, and average
Beck Anxiety Index | Week 0, Week 2, Week 4
  The BAI is a self-report questionnaire that measures the severity of anxiety. It contains 21 multiple-choice questions; each answer is scored on 0 (not at all) to 3 (severely) scale. Higher scores indicate more severe anxiety symptoms.
Beck Depression Inventory | Week 0, Week 2, Week 4
  The BDI contains 21-questions with each answer being scored on a scale value of 0 to 3 and higher scores indicating more severe depression symptoms. Scores range from minimal depression (0-13), mild depression (14-19) moderate depression (20-28) and severe depression (<29). A score of ≥ 20 indicates moderate to severe depression and the person would be excluded from participating upon completion of the baseline questionnaire.
Pittsburgh Sleep Quality Index | Week 0, Week 2, Week 4
  This is used to assess sleep quality and disturbances over a one month period. A total PSQI score of >5 indicates poor sleep quality.
Fibromyalgia 2016 | Week 0, Week 2, Week 4
  This is used to measure widespread pain and co-morbid symptoms. 2011 FM survey will be completed at pre and post sleep-restriction and post recovery period.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, Rehabilitation Science, and Athletic Training, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2025-10-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT07216417/SAP_000.pdf
  • Informed Consent Form (2025-10-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT07216417/ICF_001.pdf